CLINICAL TRIAL: NCT04760236
Title: Phase III, Multicenter, Observer-Blinded, Randomized, Active Controlled Trial to Evaluate Immune Non-Inferiority, Safety and Lot-to-Lot Consistency of OCV-S Compared to Shanchol™ in 1 to 40 Years Old Healthy Nepalese Participants
Brief Title: Immune Non-Inferiority, Safety and Lot-to-Lot Consistency of Oral Cholera Vaccine-Simplified Compared to Shanchol™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: EuBiologics Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IVI OCV-S
Record Dates: First submitted 2021-01-13; First posted 2021-02-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Cholera
MeSH Terms: conditions — Cholera | interventions — shanchol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oral Cholera Vaccine-Simplified (OCV-S) group (Lot 1) (Experimental): Participants (n=330) aged 18-40 years old will received OCV-S (Lot 1) according to 0-2 week schedule.
  Interventions: Biological: Oral Cholera Vaccine Simplified (OCV-S)
- Oral Cholera Vaccine-Simplified (OCV-S) group (Lot 2) (Experimental): Participants (n=330) aged 18-40 years old will received OCV-S (Lot 2) according to 0-2 week schedule.
  Interventions: Biological: Oral Cholera Vaccine Simplified (OCV-S)
- Oral Cholera Vaccine-Simplified (OCV-S) group (Lot 3) (Experimental): Participants (n=935) aged 1-40 years old will received OCV-S (Lot 3) according to 0-2 week schedule.
  Interventions: Biological: Oral Cholera Vaccine Simplified (OCV-S)
- Shanchol™ group (Active Comparator): Participants (n=935) aged 1-40 years old will received Shanchol™ according to 0-2 week schedule.
  Interventions: Biological: Shanchol™

INTERVENTIONS:
Biological: Oral Cholera Vaccine Simplified (OCV-S) — * Manufacturer: EuBiologics Co., Ltd.
  * Oral administration
  Arms: Oral Cholera Vaccine-Simplified (OCV-S) group (Lot 1); Oral Cholera Vaccine-Simplified (OCV-S) group (Lot 2); Oral Cholera Vaccine-Simplified (OCV-S) group (Lot 3)
Biological: Shanchol™ — * Manufacturer: Shantha Biotechnics
  * Oral administration
  Arms: Shanchol™ group

SUMMARY:
This study is to evaluate immune non-inferiority, safety and lot-to-lot consistency of OCV-S compared to Shanchol™ in 1 to 40 years old healthy Nepalese participants. The investigators hypothesize that the simplified formulation is able to induce non-inferior immunogenicity compared to licensed OCV, Shanchol™.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants 1 to 40 years of age at enrollment
* Participants/Parent(s)/Legally authorized representative (LAR) willing to provide written informed consent to participate study voluntarily
* Participants/Parent(s)/LAR who can be followed up during the study period and can comply with the study requirements

Exclusion Criteria:

* Known history of hypersensitivity reactions to other preventive vaccines
* Severe chronic diseases or medical conditions based on the medical judgment of the investigator. In particular, a participant with a) chronic infection such as tuberculosis, or sequel of poliomyelitis, b) known history of immune function disorders, c) chronic use of systemic steroids (>2 mg/kg/day or >20 mg/day prednisone equivalent for periods exceeding 10 days)/cytotoxic drugs/immunosuppressants within past 6 weeks, d) active malignancy with the exception of adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I cancer from which the participant is currently in complete remission, or any other cancer from which the participant has been disease-free for 5 years, e) Congestive heart failure, f) myocardial infarction within the previous 6 months, g) known HIV-infected patients, h) neurological and/or psychiatric disorder, or i) known history of uncontrolled coagulopathy or blood disorders
* Participant who planned to or has received other vaccines from 1 month prior to test vaccination excluding a public health vaccination campaign due to an outbreak
* Participant concomitantly enrolled or scheduled to be enrolled in another trial
* Receipt of blood or blood-derived products in the past 3 months
* Participant who has previously received a cholera vaccine
* Any female participant who is lactating, pregnant or planning for pregnancy during study period
* Participants planning to move from the study area before the end of study period
* Employees or the family members of the OCV-S study sites

Temporary Contraindication:

Should a participant have one of the conditions/situations listed below, the Investigator will postpone primary or subsequent vaccination until the condition/situation is resolved.

* Febrile illness (axillary temperature ≥ 37.5°C) or moderate or severe acute illness/infection on the day of vaccination or planned vaccination, according to Investigator's judgment.
* Gastrointestinal symptoms including nausea, vomiting, or decreased appetite within 24 hours prior to study initiation.
* Administration of antidiarrheal drugs or antibiotics to treat diarrhea or abdominal pain lasting 2 weeks or longer within 6 months prior to study initiation
* Diarrhea occurring up to 1 week within 6 months prior to study initiation.

  * Lactation: Breastfeeding women will not be enrolled. Should a female participant decide to breastfeed during the vaccination period, she will be excluded from further vaccination, but will be followed for safety until the end of the study
  * Pregnancy Test is necessary for all married female participants of childbearing age.

Ages: 1 Year to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2530 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Immune non-inferiority of OCV-S compared to Shanchol™ (i.e., one lot of OCV-S) as measured by seroconversion rates for all ages | 2 weeks after second dose of either OCV-S (i.e., one lot of OCV-S) or Shanchol™
  Proportion of participants showing seroconversion of vibriocidal titers against Vibrio cholerae O1 Inaba and O1 Ogawa 2 weeks after second dose of either OCV-S (i.e., one lot of OCV-S) or Shanchol™ for all ages
Vaccine Safety profile | As in Description
  Frequency of solicited adverse events within 7 days post vaccination, unsolicited adverse events within 28 days post vaccination, Serious Adverse Events (SAEs) after each dose during the entire study period in all ages and in each age stratum

SECONDARY OUTCOMES:
Immune non-inferiority of OCV-S compared to Shanchol™ (i.e., one lot of OCV-S) as measured by GMT for all ages | 2 weeks after second dose of either OCV-S (i.e., one lot of OCV-S) or Shanchol™
  Geometric Mean Titer (GMT) of vibriocidal antibodies against Vibrio cholerae O1 Inaba and Ogawa 2 weeks after second dose of either OCV-S (i.e., one lot of OCV-S) or Shanchol™ for all ages
Immune non-inferiority of OCV-S compared to Shanchol™ (i.e., one lot of OCV-S) as measured by seroconversion rate in each age stratum | 2 weeks after second dose of either OCV-S (i.e., one lot of OCV-S) or Shanchol™
  Proportion of participants showing seroconversion against Vibrio cholerae O1 Inaba and Ogawa 2 weeks after second dose of either OCV-S (i.e., one lot of OCV-S) or Shanchol™ in each age stratum
Immune non-inferiority of OCV-S compared to Shanchol™ (i.e., one lot of OCV-S) as measured by GMT in each age stratum | 2 weeks after second dose of either OCV-S (i.e., one lot of OCV-S) or Shanchol™
  Geometric Mean Titer of vibriocidal antibodies against Vibrio cholerae O1 Inaba and Ogawa 2 weeks after second dose of either OCV-S (i.e., one lot of OCV-S) or Shanchol™ in each age stratum
The equivalence of immunogenicity in 3 lots as measured by GMT | 2 weeks after second dose of either OCV-S (i.e., one lot of OCV-S) or Shanchol™
  Geometric Mean Titer of vibriocidal antibodies against Vibrio cholerae O1 Inaba and Ogawa 2 weeks after second dose of 3 lots of OCV-S in adults

OTHER OUTCOMES:
The equivalence of immunogenicity in 3 lots as measured by seroconversion rates | 2 weeks after second dose of either OCV-S (i.e., one lot of OCV-S) or Shanchol™
  Proportion of participants showing seroconversion of vibriocidal titers against Vibrio cholerae O1 Inaba and Ogawa 2 weeks after second dose of 3 lots of OCV-S in adults
Vibriocidal antibody responses | 2 weeks after first dose of either OCV-S (i.e., one lot of OCV-S) or Shanchol™
  Seroconversion rate and GMT of vibriocidal antibody responses 2 weeks after first dose for all ages and for each age stratum

CONTACTS AND LOCATIONS:
Overall Officials: Julia Lynch, MD, Principal Investigator — International Vaccine Institution
Locations (4):
- Nepal (4):
  - Nepalgunj medical college, Bānke, City- Nepalgunj
  - B.P.Koirala Institute of Health Sciences, Rautahat, Dharan
  - Dhulikhel Hospital, Kavre, Dhulikhel
  - Kanti Children's Hospital, Kathmandu, Sukedhara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song KR, Chapagain RH, Tamrakar D, Shrestha R, Kanodia P, Chaudhary S, Wartel TA, Yang JS, Kim DR, Lee J, Park EL, Cho H, Lee J, Thaisrivichai P, Vemula S, Kim BM, Gupta B, Saluja T, Pansuriya RK, Ganapathy R, Baik YO, Lee YJ, Jeon S, Park Y, Her HL, Park Y, Lynch JA. Safety and immunogenicity of the Euvichol-S oral cholera vaccine for prevention of Vibrio cholerae O1 infection in Nepal: an observer-blind, active-controlled, randomised, non-inferiority, phase 3 trial. Lancet Glob Health. 2024 May;12(5):e826-e837. doi: 10.1016/S2214-109X(24)00059-7. PMID 38614631